CLINICAL TRIAL: NCT04395638
Title: Replenishing and Maintaining Vitamin D Status in Deficient Older Adults in Residential Care Facilities in Northern Ireland
Brief Title: Replenishing and Maintaining Vitamin D Status in Older Adults in Residential Care Facilities in NI
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 study status being reviewed on an ongoing basis.
Sponsor: University of Ulster (Other)
Collaborators: Western Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/NI/0031
Record Dates: First submitted 2020-05-11; First posted 2020-05-20 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Deficiency; Bone Health; Generic Health Relevance; Musculoskeletal Health; Intervention
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly Vitamin D group (Experimental)
  Interventions: Dietary Supplement: 20,000IU Vitamin D3 per week for 8 weeks
- Daily Vitamin D group (Experimental)
  Interventions: Dietary Supplement: 3200IU Vitamin D3 per day for 8 weeks

INTERVENTIONS:
Dietary Supplement: 3200IU Vitamin D3 per day for 8 weeks — 3200IU Vitamin D3 per day for 8 weeks
  Arms: Daily Vitamin D group
Dietary Supplement: 20,000IU Vitamin D3 per week for 8 weeks — 20,000IU Vitamin D3 per week for 8 weeks
  Arms: Weekly Vitamin D group

SUMMARY:
The vitamin D status of older adults in residential care facilities in Northern Ireland (NI) is currently unknown. An observation study is currently being carried out by Ulster University and the Western Health & Social Care Trust (WHSCT) to provide data on the prevalence of vitamin-D deficiency among older adults within residential care facilities in NI. It is expected that some 40% of the cohort will be deficient in vitamin D and will require immediate replenishment of vitamin D status. Therefore, as a follow up to the observational study, an intervention study will be conducted, where participants identified as vitamin D deficient (25(OH)D) status <30nmol/L (cut-off currently used by the WHSCT will be re-contacted and provided with a vitamin D supplement. The aim of this study is to investigate the dose and duration of vitamin D supplementation that is required to replenish and maintain vitamin D status in older adults with vitamin D deficiency within residential care facilities. Participants will be randomly assigned to receive one of two supplementation regimes: 3200IU/day vitamin D3 or 20,000IU/week vitamin D3. Blood samples (no more than 20ml per appointment) will be taken at 4 different time points: week 0, week 2, week 4 and week 8. These two doses are routinely used in clinical practice for remedial supplementation of vitamin D and have been chosen based upon their availability from manufacturers of vitamin D supplements. Also, albeit these doses are currently routinely used to replenish vitamin D status little is known on how effective they are and how soon vitamin D status is optimised. Clinicians can only administer medication for the management of osteoporosis (e.g. bisphosphonates) once vitamin D status is optimised. Therefore, measurements will be taken every two weeks to establish response to the remedial supplementation. This project provides a unique opportunity to monitor the replenishment and maintenance of vitamin D status following remedial supplementation more regularly (at weeks 0,2,4,8) than would be done under standard National Health Service care. This does and duration of vitamin D required to replenish vitamin D deficiency in older adults is currently ambiguous within the literature and clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Currently residing (≥1 month) within residential care facilities in Northern Ireland and who have previously undertaken the observation study (full title: A cross-sectional analysis of vitamin D status and bone health of older adults within residential care facilities in Northern Ireland) and have been identified as vitamin D deficient.

Exclusion Criteria:

* Participants will be excluded from the study if by the judgement of the consultant rheumatologist that they have very abnormal bone or vitamin D metabolism due to conditions such as end stage renal failure or bone metastases.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Vitamin D status | Change between baseline (week 0 pre-intervention) and weeks 2, 4, 8 post-intervention
  Plasma 25(OH)D status analysis by Liquid Chromatography / Mass Spec (LC/MS)

SECONDARY OUTCOMES:
Osteocalcin concentration | Change between baseline (week 0 pre-intervention) and weeks 2, 4, 8 post-intervention
  Bone turnover marker
Bone-specific alkaline phosphatase concentration | Change between baseline (week 0 pre-intervention) and weeks 2, 4, 8 post-intervention
  Bone turnover marker

CONTACTS AND LOCATIONS:
Locations (1):
- Western Health and Social Care Trust Care Home facilities, Londonderry, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No